CLINICAL TRIAL: NCT04512781
Title: Clinical Efficacy in Relief of Dyspnea by HVNI: Evaluation of New Cannulae Designs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vapotherm, Inc. (Industry)
Collaborators: VA Pittsburgh Healthcare System (U.S. Federal Agency); Erlanger Baroness Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RP-VTPF2018002Sci
Record Dates: First submitted 2020-08-06; First posted 2020-08-14 (Actual); Results first posted 2024-02-23 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Dyspnea; Hypercapnia; Respiratory Insufficiency
MeSH Terms: conditions — Dyspnea; Hypercapnia; Respiratory Insufficiency

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Conventional Legacy Cannula Design (Control) - Prosoft Cannula - Unicorn Cannula (Experimental): During this session, patients will be placed on HVNI therapy with an appropriately fitted Vapotherm conventional legacy cannula. Physiologic and ventilation parameters will be recorded.
  Patients will be randomly assigned to Prosoft or Unicorn cannula testing groups. Physiologic and ventilation parameters will be recorded.
  Interventions: Device: Control Cannula - Prosoft Cannula - Unicorn Cannula
- Conventional Legacy Cannula Design (Control) - Unicorn Cannula - Prosoft Cannula (Experimental): During this session, patients will be placed on HVNI therapy with an appropriately fitted Vapotherm conventional legacy cannula. Physiologic and ventilation parameters will be recorded.
  Patients will be randomly assigned to Prosoft or Unicorn cannula testing groups. Physiologic and ventilation parameters will be recorded.
  Interventions: Device: Control Cannula - Unicorn Cannula - Prosoft Cannula

INTERVENTIONS:
Device: Control Cannula - Prosoft Cannula - Unicorn Cannula — The purpose of this intervention is to evaluate the efficacy of a conventional legacy cannula design to provide targeted relief of dyspnea. The purpose of this intervention is to evaluate the efficacy of a next generation cannula to provide relief of dyspnea.
  Arms: Conventional Legacy Cannula Design (Control) - Prosoft Cannula - Unicorn Cannula
Device: Control Cannula - Unicorn Cannula - Prosoft Cannula — The purpose of this intervention is to evaluate the efficacy of a conventional legacy cannula design to provide targeted relief of dyspnea. The purpose of this intervention is to evaluate the efficacy of a next generation cannula to provide relief of dyspnea.
  Arms: Conventional Legacy Cannula Design (Control) - Unicorn Cannula - Prosoft Cannula

SUMMARY:
This study will evaluate the ability of High Velocity Nasal Insufflation [HVNI] next generation nasal cannula designs to effect ventilation and related physiological responses relative to the conventional legacy cannula design.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the ability of HVNI next generation nasal cannula designs to effect ventilation and related physiological responses relative to the current cannula design, with which there are published clinical outcomes data. It is hypothesized that next generation nasal cannula designs (Prosoft and Unicorn) will be comparable at relieving patient dyspnea while on HVNI, when compared to the conventional (Legacy) cannula.

ELIGIBILITY:
Inclusion Criteria:

* Adults, 18 years or older
* Demonstrated severe dyspnea at baseline (Borg Rated Perceived Dyspnea [RPD] (scale 0-10) of 3 or higher)
* Severe baseline hypercarbia/hypercapnia of 50 mmHg or higher as measured by TcPCo2 or arterial or venous blood gas

Exclusion Criteria:

* Patient has unstable cardiovascular condition
* Significant unilateral or bilateral nasal occlusion
* Vigorous physical activity should not be performed within 2 hours of testing
* Inability to provide informed consent
* Pregnancy
* Known contraindication to perform steps of the protocol
* Absence of spontaneous respiration or known contraindication to HVNI
* Inability to use nasal cannula and HVNI therapy
* Agitation or uncooperativeness
* Determined by the clinician to be sufficiently unstable or unsuitable for this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2022-06-07 (Actual); Study Completion 2022-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles W Atwood, MD, FCCP, Principal Investigator — VA Pittsburgh Healthcare System; Jigme M Sethi, MD, FCCP, Principal Investigator — Erlanger Baroness Hospital
Locations (2):
- United States (2):
  - VA Pittsburgh Healthcare System, Pittsburgh, Pennsylvania
  - Erlanger Baroness Hospital, Chattanooga, Tennessee

RESULTS

PARTICIPANT FLOW:
Groups:
- Conventional Legacy Cannula Design (Control) - Prosoft Cannula - Unicorn Cannula: Conventional Legacy Cannula Design (Control) first for 40 min, then Prosoft Cannula for 40min - then Unicorn Cannula for 40 min")
- Conventional Legacy Cannula Design (Control) - Unicorn Cannula - Prosoft Cannula: Conventional Legacy Cannula Design (Control) first for 40 min, then Unicorn Cannula for 40min - then Prosoft Cannula for 40 min")
Period: Overall Study
Arm/Group | Conventional Legacy Cannula Design (Control) - Prosoft Cannula - Unicorn Cannula | Conventional Legacy Cannula Design (Control) - Unicorn Cannula - Prosoft Cannula
Started | 15 | 11
Completed | 15 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Conventional Legacy Cannula Design (Control) - Prosoft Cannula - Unicorn Cannula: During this session, patients will be placed on HVNI therapy with an appropriately fitted Vapotherm conventional legacy cannula. Physiologic and ventilation parameters were recorded.
  Patients were assigned to go on the Prosoft Cannula second. Physiologic and ventilation parameters were recorded.
  Patients were assigned to go on the Unicorn Cannula third. Physiologic and ventilation parameters were recorded
- Conventional Legacy Cannula Design (Control) - Unicorn Cannula - Prosoft Cannula: During this session, patients will be placed on HVNI therapy with an appropriately fitted Vapotherm conventional legacy cannula. Physiologic and ventilation parameters were recorded.
  Patients were assigned to go on the Unicorn Cannula second. Physiologic and ventilation parameters were recorded.
  Patients were assigned to go on the Prosoft Cannula third. Physiologic and ventilation parameters were recorded.
- Total: Total of all reporting groups
Arm/Group | Conventional Legacy Cannula Design (Control) - Prosoft Cannula - Unicorn Cannula | Conventional Legacy Cannula Design (Control) - Unicorn Cannula - Prosoft Cannula | Total
Number analyzed (Participants) | 15 | 11 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 10 | 9 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 11 | 7 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 10 | 23
  Unknown or Not Reported | 2 | 1 | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 2 | 7
  White | 9 | 9 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
height [Median (Full Range); unit: m] — There was a median calculated for all the participants, with a range of 1.7m to 1.80m
  m | 1.78 [1.7 to 1.8] | 1.72 [1.7 to 1.8] | 1.77 [1.7 to 1.8]
Weight [Median (Full Range); unit: kg] — a median for weight was calculated for all the participants, with a range of 82kg to 128kg
  kg | 108.8 [82 to 128] | 86.18 [82 to 128] | 91 [82 to 128]

OUTCOME MEASURES:

1. Primary Outcome: Patient Vital Signs -- Rated Perceived Dyspnea (RPD)
Description: Patient's subjective assessment of their dyspnea, rated as a modified Borg score on a scale from 0 to 10. Higher scores indicate a worse outcome.
Time Frame: This was collected at the end of each phase, for a total of three phases over the course of the study (2 hours 15 min)
Measure: Median (95% Confidence Interval); unit: units on a scale
Groups:
- Legacy Cannula: During this session, participants completed the entire study intervention while wearing the Legacy Cannula. Physiologic and ventilation parameters were recorded.
- Prosoft Cannula: During this session, participants completed the entire study intervention while wearing the Prosoft Cannula. Physiologic and ventilation parameters were recorded.
- Unicorn Cannula: During this session, participants completed the entire study intervention while wearing the Unicorn Cannula. Physiologic and ventilation parameters were recorded.
Arm/Group | Legacy Cannula | Prosoft Cannula | Unicorn Cannula
Number analyzed (Participants) | 26 | 26 | 26
units on a scale | 3 [3 to 3] | 2.5 [2 to 3] | 2.5 [2 to 3]

2. Secondary Outcome: Patient Vital Signs - Heart Rate [HR]
Description: Heart Rate (HR) The number of beats per minute.
Time Frame: This was collected at the end of each phase, for a total of three phases over the course of the study (2 hours 15 min)
Measure: Median (95% Confidence Interval); unit: Beats per minute
Arm/Group | Legacy Cannula | Prosoft Cannula | Unicorn Cannula
Number analyzed (Participants) | 26 | 26 | 26
Beats per minute | 78 [73 to 85] | 74 [71 to 79] | 76 [69 to 80]

3. Secondary Outcome: Patient Vital Signs - Respiratory Rate [RR]
Description: Respiratory rate, measured in breaths per minute (brpm)
Time Frame: This was collected at the end of each phase, for a total of three phases over the course of the study (2 hours 15 min)
Measure: Median (95% Confidence Interval); unit: BRPM
Arm/Group | Legacy Cannula | Prosoft Cannula | Unicorn Cannula
Number analyzed (Participants) | 26 | 26 | 26
BRPM | 16 [15 to 20] | 18 [14 to 20] | 16 [14 to 19]

4. Secondary Outcome: Patient Vital Signs - Blood Pressure [BP]
Description: Blood pressure (systolic) measured in mmHg
Time Frame: This was collected at the end of each phase, for a total of three phases over the course of the study (2 hours 15 min)
Measure: Median (95% Confidence Interval); unit: mmHg
Arm/Group | Legacy Cannula | Prosoft Cannula | Unicorn Cannula
Number analyzed (Participants) | 26 | 26 | 26
mmHg
  Systolic | 126 [119.25 to 132.75] | 126 [119.52 to 132.48] | 123 [114.62 to 131.38]
  Diastolic | 71 [66.41 to 75.60] | 71 [66.75 to 75.25] | 69 [64.80 to 73.20]

5. Secondary Outcome: Patient Vital Signs - Arterial Oxygen Saturation [SpO2]
Description: SpO2 measured as percentage of oxygen saturation (%)
Time Frame: This was collected at the end of each phase, for a total of three phases over the course of the study (2 hours 15 min)
Measure: Median (95% Confidence Interval); unit: percentage of oxygen saturation
Arm/Group | Legacy Cannula | Prosoft Cannula | Unicorn Cannula
Number analyzed (Participants) | 26 | 26 | 26
percentage of oxygen saturation | 95 [93 to 97] | 95 [93 to 96] | 95 [93 to 96]

6. Secondary Outcome: Patient Vital Signs - Transcutaneous CO2 [TcPCO2]
Description: TcPCO2 measured as percentage of CO2 (%)
Time Frame: This was collected at the end of each phase, for a total of three phases over the course of the study (2 hours 15 min)
Measure: Median (95% Confidence Interval); unit: percentage of CO2
Arm/Group | Legacy Cannula | Prosoft Cannula | Unicorn Cannula
Number analyzed (Participants) | 26 | 26 | 26
percentage of CO2 | 53.8 [46 to 60] | 50.7 [46 to 57] | 50.3 [45 to 56]

7. Other Pre Specified Outcome: Clinician Perception Score - Frequency of Technical/Clinical Difficulties
Description: Clinician's subjective assessment of the frequency of technical or clinical issues during the the test, rated as units on a visual analog scale from 0 to 100. Lower scores indicate a better outcome.
Time Frame: This was collected at the end of each phase, for a total of three phases over the course of the study (2 hours 15 min)
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Clinician Perception Score - Patient Comfort/Tolerance
Description: Clinician's subjective assessment of the patient's comfort and tolerance of therapy during the the test, rated as units on a visual analog scale from 0 to 100. Lower scores indicate a better outcome.
Time Frame: Through study completion, an average of 3 hours
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Clinician Perception Score - Ease of Use
Description: Clinician's subjective assessment of the ease of use of therapy during the the test, rated as units on a visual analog scale from 0 to 100. Lower scores indicate a better outcome.
Time Frame: Through study completion, an average of 3 hours
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Clinician Perception Score - Monitoring & Support for Therapy
Description: Clinician's subjective assessment of the level of monitoring and support for therapy required during the the test, rated as units on a visual analog scale from 0 to 100. Lower scores indicate a better outcome.
Time Frame: Through study completion, an average of 3 hours
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Clinician Perception Score - Expected/Perceived Patient Outcomes
Description: Clinician's subjective assessment of the expected and perceived patient outcomes as a result of therapy following testing, rated as units on a visual analog scale from 0 to 100. Lower scores indicate a better outcome.
Time Frame: Through study completion, an average of 3 hours
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Patient Perception Score - Relief of Symptoms
Description: Patient's subjective assessment of relief of their symptoms while on therapy, rated as units on a visual analog scale from 0 to 100. Lower scores indicate a better outcome.
Time Frame: Through study completion, an average of 3 hours
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Patient Perception Score - Comfort/Tolerance of Therapy
Description: Patient's subjective assessment of their comfort and tolerance of therapy during the the test, rated as units on a visual analog scale from 0 to 100. Lower scores indicate a better outcome.
Time Frame: Through study completion, an average of 3 hours
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Adverse Event reporting and collection was done over the duration of the trial, approximately 2 hours and 15 min.
Description: Any untoward or unfavorable medical occurrence in a participant, including any abnormal sign (for example, abnormal physical exam or laboratory finding), symptom, or disease, temporally associated with the participant's participation in the research, whether or not considered related to the participant's participation in the research.
Arm/Group | Legacy Cannula | Prosoft Cannula | Unicorn Cannula
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/26 | 0/26
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 0/26 | 0/26 | 0/26

LIMITATIONS AND CAVEATS:
Small sample size and very specific scope of measuring RPD. Study was done during COVID pandemic. Screening efforts restricted to the ICU. Measurements were done with newer cannulas followed by legacy cannula. The study was non blinded. Patients may not have been aware of the difference between the legacy and the Prosoft cannula.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-06-10): https://cdn.clinicaltrials.gov/large-docs/81/NCT04512781/Prot_SAP_000.pdf